CLINICAL TRIAL: NCT00577837
Title: Active-controlled, Double-blind, Randomized, Sequential Escalating Dose Study to Assess Safety, Pharmacokinetics and Efficacy of 100, 150, and 200 mg Oral Risedronate Administered Monthly in Postmenopausal Women With Low Bone Mineral Density
Brief Title: Safety, Pharmacokinetics, and Efficacy of 100, 150, and 200 mg Risedronate Administered to Women With Low BMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003134; HMR4003K/2001
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Postmenopausal
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 5 mg risedronate, once daily for 6 months
  Interventions: Drug: risedronate
- 2 (Experimental): 100 mg risedronate, once a month for 6 months
  Interventions: Drug: risedronate
- 3 (Experimental): 150 mg risedronate, once a month for 6 months
  Interventions: Drug: risedronate
- 4 (Experimental): 200 mg risedronate, once a month for 6 months
  Interventions: Drug: experimental

INTERVENTIONS:
Drug: risedronate — tablet, 5 mg risedronate daily for 6 months
  Arms: 1
Drug: risedronate — tablet, 100 mg risedronate monthly for 6 months
  Arms: 2
Drug: risedronate — tablet, 150 mg risedronate monthly for 6 months
  Arms: 3
Drug: experimental — tablet, 200 mg risedronate monthly for 6 months
  Arms: 4

SUMMARY:
A Multi-center, Active-controlled (5 mg daily risedronate), Double-blind, Randomized, Sequential Escalating Dose Study to Assess Safety, Pharmacokinetics and Efficacy of 100, 150, and 200 mg Oral Risedronate Administered Monthly for Six Months in Postmenopausal Women with Low Bone Mineral Density.

ELIGIBILITY:
Inclusion Criteria:

* be postmenopausal 5 years based on medical history; follicle stimulating hormone and estradiol will be evaluated for any patient less than 65 years of age, who has undergone hysterectomy without bilateral oophorectomy, to ensure the patient is postmenopausal

Exclusion Criteria:

* use of any of the following medications within 3 months of starting study drug or use of any of the following medications for more than 1 month at any time within 6 months prior to starting study drug:

  * oral or parenteral glucocorticoids (5 mg prednisone or equivalent per day)
  * anabolic steroids
  * estrogen, raloxifene or estrogen-related drugs, eg, tamoxifen, tibolone, (except for low dose vaginal creams, tablets or insertable estrogen ring
  * progestogen
  * calcitonin
  * vitamin D supplements (greater than 800 IU per day)
  * calcitriol, calcidiol, or alfacalcidol
  * any bisphosphonate
  * fluoride (10 mg per day)
  * strontium and other bone active agents
  * parathyroid hormone
  * heparin, warfarin, and other similar anticoagulants

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of 3 once-monthly dosing regimens of risedronate, 100 mg, 150 mg and 200 mg, compared to a once-daily dosing regimen, 5 mg, as assessed by clinical laboratory values and adverse event (AE) profiles | 6 months

SECONDARY OUTCOMES:
Evaluate the efficacy of 3 once-monthly dosing regimens or risedronate compared to a once-daily dosing regimen and to evaluate the PK/PD of monthly and daily dose regimens | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Beary, MD, Study Director — Procter and Gamble
Locations (14):
- United States (4):
  - Research Site, Daytona Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Shawnee Mission, Kansas
  - Research Site, San Antonio, Texas
- Canada (3):
  - Research Site, Hamilton, Ontario
  - Research Facility, Montreal, Quebec
  - Research Facility, Sainte-Foy, Quebec
- Research Facility, Zagreb, Croatia
- Netherlands (2):
  - Research Facility, Amsterdam
  - Research Facility, Leiden
- Poland (4):
  - Research Facility, Bialystok
  - Research Site, Lublin
  - Research Site, Warsaw
  - Research Site, Wroclaw